CLINICAL TRIAL: NCT07131631
Title: Secondary Mitral Regurgitation Treatment With MitraClip and Assessment by Cardiac Magnetic Resonance
Acronym: SMARTER-CMR
Status: Recruiting | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1807968
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure and Reduced Ejection Fraction; Functional Mitral Regurgitation
Keywords: heart failure; reduced ejection fraction; functional mitral regurgitation
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 group undergoing guideline directed TEER with FDA approved MitraClip: Cohort will undergo a clinically indicated baseline CMR study with contrast up to 90 days before TEER procedure. Quality of life questionnaire will also be completed. At 6 months, individuals will return to the clinic to repeat quality of life questionnaires, the CMR study and a transthoracic echocardiogram.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Clinically indicated baseline CMR study with contrast up to 90 days before TEER procedure, including KCCQ questionnaire. At 6 months, participants will return for repeat of KCCQ, CMR study and a transthoracic echocardiogram. Blood samples, done as standard clinical care for hemotocrit for ECV calculation, will be obtained.
  Other Names: Transthoracic echocardiogram

SUMMARY:
This is a multi-center, prospective, observational study designed to evaluate the impact of LV myocardial fibrosis extent assessed by CMR on LV reverse remodeling and clinical outcomes post TEER. The target sample will be up to 125 patients enrolled to achieve 100 evaluable at 6 months of follow-up. Enrollment will occur at up to eight centers.

DETAILED DESCRIPTION:
Patients undergoing guideline-directed TEER with FDA-approved MitraClip at the participating centers will be screened and recruited for study participation. After informed consent is obtained, patients will undergo a clinically-indicated baseline CMR study with gadolinium up to 90 days before TEER procedure. In addition, a quality-of-life surveillance questionnaire (KCCQ) will be completed at the same baseline visit.

Six months after TEER patients will return to clinic to repeat the quality of life surveillance questionnaire (KCCQ), the CMR study and a transthoracic echocardiogram. The 6-month CMR study and echocardiogram should be completed on the same day or no greater than 30 days apart if the same day is not feasible. Blood samples will be collected on the day of the CMR to provide the hematocrit for ECV calculation. These samples are done as standard clinical care.

Electronic Health Records (EHR) will be reviewed and phone contact performed yearly for up to three years after TEER to evaluate clinical outcomes (heart failure hospitalization, outpatient use of intravenous inotropes, LVAD implant, heart transplant, or death).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) with heart failure and reduced ejection fraction (LVEF < 50% defined by echocardiography), medically and device-optimized according to guidelines, with significant FMR undergoing TEER with FDA-approved MitraClip device (Abbott Structural, USA)

Exclusion Criteria:

1. Concomitant PCI and TEER
2. Congenital heart disease
3. Stage D heart failure
4. Uncontrolled atrial fibrillation
5. Pregnancy
6. > moderate tricuspid regurgitation
7. >moderate aortic regurgitation or stenosis
8. Contraindications or unable to undergo CMR
9. Prior mitral valve repair or replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing guideline-directed TEER with FDA-approved MitraClip at the participating centers will be screened and recruited for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Estimate the association between LV myocardial fibrosis by CMR late gadolinium enhancement imaging before TEER with LV reverse remodeling. | From enrollment to the end of 6 months
  change in LV end-diastolic volume index [LVEDVi] 6 months after TEER

SECONDARY OUTCOMES:
Estimate the association of the ratio between CMR-based mitral regurgitant volume (RegVol) and LV end-diastolic volume (LVEDV)-RegVol/LVEDV-with LV reverse remodeling; | Enrollment to the end of 6 months
  Reg/Vol and LVEDV with LV reverse remodeling
Evaluate the interaction between CMR-based mitral regurgitation quantification (RegVol and regurgitant fraction) with LV myocardial fibrosis extent, and its association with LV reverse remodeling | Enrollment to the end of 6 months
  RegVol and regurgitant fraction with LV myocardial fibrosis extent
Estimate the association between LV extracellular volume (ECV) by CMR T1 mapping before TEER with LV reverse remodeling | Enrollment to the end of 6 months
  ECV before TEER with LV reverse remodeling
Estimate the association of LV myocardial fibrosis extent and a combined endpoint including all-cause death, heart failure hospitalization, cardiac transplant and LVAD implant; | Enrollment to the end of 6 months
  LV myocardial fibrosis and endpoint data points (all cause death, heart failure hospitalization, cardiac transplant and LVAD implant)
Estimate the association of LV myocardial fibrosis extent and the change in quality-of-life (Kansas City Cardiomyopathy Questionnaire [KCCQ]) post TEER | Enrollment to the end of 6 months
  LV myocardial extent and % of change in quality of life KCCQ
Estimate the intermodality agreement of residual MR between 3D echo and CMR at 6 months post-TEER | Enrollment through 6 months
  Intermodality agreement of residential agreement in echo and CMR

CONTACTS AND LOCATIONS:
Overall Officials: João Cavalcante, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (6):
- United States (5):
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - The Christ Hospital Health Network, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Only de-identified data may be shared/published.